CLINICAL TRIAL: NCT00067613
Title: Randomized Controlled Trial of Benchmarking to Reduce Bronchopulmonary Dysplasia to Reduce Bronchopulmonary Dysplasia
Brief Title: Benchmarking Initiative to Reduce Bronchopulmonary Dysplasia
Acronym: Benchmarking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Michele C. Walsh, Lead Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NICHD-NRN-0025; U10HD034216 (NIH); U10HD021364 (NIH); U10HD027853 (NIH); U10HD027851 (NIH); U01HD036790 (NIH); U10HD027856 (NIH); U10HD021397 (NIH); U10HD027881 (NIH); U10HD027880 (NIH); U10HD021415 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); U10HD034167 (NIH); U10HD027904 (NIH); M01RR008084 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR000070 (NIH); M01RR006022 (NIH); M01RR002635 (NIH); M01RR002172 (NIH); M01RR001032 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-26 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Bronchopulmonary Dysplasia (BPD)
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity; Mechanical ventilation; Benchmarking; Chronic Lung Disease (CLD)
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Clinical sites randomized to intervention will receive training in the benchmarking BPD management methods identified at the Benchmark sites.
  Interventions: Other: Benchmarking Management Practices
- Control (Placebo Comparator): Clinical sites randomized to Control will continue with their normal management practices for BPD.
  Interventions: Other: Standard Management Practices

INTERVENTIONS:
Other: Benchmarking Management Practices — The Benchmarking intervention included:
  1. Data feedback: Using existing data from the NRN Generic Database and Key Care Practices Survey at their NICU to collect data on the perceptions of care.
  2. Training in Continuous Quality Improvement (CQI) Techniques
  3. Review of best existing evidence
  4. Site visits to the Centers with the Lowest Rates of BPD
  5. Selection of Practices to change: Each site team selected practices for modification at their own center
  Arms: Intervention
Other: Standard Management Practices — Centers assigned to the control group continued to receive routine information on their own center's outcomes, and all information routinely supplied within the NRN. Control centers did not participate in organized discussions of the interventions applied within the Benchmarking centers. At the completion of the study, Control Centers were offered a workshop on the Benchmarking techniques.
  Arms: Control

SUMMARY:
This study tested whether Neonatal Intensive Care Unit (NICU) teams trained in benchmarking -- comparing care practices between different NICUs to see which practices prevent bronchopulmonary dysplasia (BPD) -- and quality improvement would change practices and improve rates of survival without BPD in inborn neonates with birth weights of <1250 grams. Benchmarking is a method involving detailed comparisons of processes between similar organizations. For this study, three NRN centers with the lowest rates of BPD have been identified as Benchmark centers. During a 6-month pre-intervention period, details of care practices and management style at these centers were carefully assessed. Based on practices at these Benchmarking sites, we developed a quality improvement program. For this study, 14 other NRN sites were randomized to either implement the benchmarking intervention (intervention sites) or continue with their usual care practices (control sites). After the 1-year intervention period, we compared changes in the rate of survival without BPD at 36 weeks corrected age between the intervention and control sites.

DETAILED DESCRIPTION:
In 1998, 55% of Very Low Birth Weight (VBLW) infants (those born at <1,250g) born at centers in the National Institute of Child Health and Human Development (NICHD) Neonatal Research Network (NRN) either died or developed BPD.

Previous studies within the NICHD Neonatal Research Network showed substantial differences in the incidence of BPD between centers. These differences were not explained by birth weight, gestational age, race, frequency of antenatal steroid use, or incidence of respiratory distress syndrome. Practice differences may contribute to BPD incidence variation. This study evaluated the efficacy of a Benchmarking Initiative to modify clinical care practices and decrease incidence of BPD in VLBW infants.

This study tested whether Neonatal Intensive Care Unit (NICU) teams trained in benchmarking -- comparing care practices between different NICUs to see which practices prevent bronchopulmonary dysplasia (BPD) -- and quality improvement would change practices and improve rates of survival without BPD in inborn neonates with birth weights of <1250 grams. Benchmarking is a method involving detailed comparisons of processes between similar organizations. For this study, three NRN centers with the lowest rates of BPD have been identified as Benchmark centers. During a 6-month pre-intervention period, details of care practices and management style at these centers were carefully assessed. Based on practices at these Benchmarking sites, we developed a quality improvement program. For this study, 14 other NRN sites were randomized to either implement the benchmarking intervention (intervention sites) or continue with their usual care practices (control sites). After the 1-year intervention period, we compared changes in the rate of survival without BPD at 36 weeks corrected age between the intervention and control sites.

ELIGIBILITY:
Inclusion Criteria

* Infants 501-1,249g birthweight
* Registered in a participating site

Exclusion Criteria

* Diagnosed with a syndrome as defined by the Neonatal Research Network's Generic Database Study

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4095 (Actual)
Dates: Start 2001-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Survival without BPD | 36 weeks of life

SECONDARY OUTCOMES:
Bronchopulmonary Dysplasia | 36 weeks of life

CONTACTS AND LOCATIONS:
Overall Officials: Michele C. Walsh, MD, Study Director — Case Western Reserve University, Rainbow Babies & Children's Hospital; William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Shahnaz Duara, MD, Principal Investigator — University of Miami; Barbara J. Stoll, MD, Principal Investigator — Emory University; James A. Lemons, MD, Principal Investigator — Indiana University; David K. Stevenson, MD, Principal Investigator — Stanford University; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Abbot R. Laptook, MD, Principal Investigator — University of Texas Southwestern Medical Center; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Jon E. Tyson, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; W. Kenneth Poole, PhD, Principal Investigator — RTI International
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Bhandari V, Finer NN, Ehrenkranz RA, Saha S, Das A, Walsh MC, Engle WA, VanMeurs KP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Synchronized nasal intermittent positive-pressure ventilation and neonatal outcomes. Pediatrics. 2009 Aug;124(2):517-26. doi: 10.1542/peds.2008-1302. Epub 2009 Jul 27. PMID 19651577
- [Result] Laptook AR, Salhab W, Allen J, Saha S, Walsh M. Pulse oximetry in very low birth weight infants: can oxygen saturation be maintained in the desired range? J Perinatol. 2006 Jun;26(6):337-41. doi: 10.1038/sj.jp.7211500. PMID 16598294
- [Result] Shankaran S, Langer JC, Kazzi SN, Laptook AR, Walsh M; National Institute of Child Health and Human Development Neonatal Research Network. Cumulative index of exposure to hypocarbia and hyperoxia as risk factors for periventricular leukomalacia in low birth weight infants. Pediatrics. 2006 Oct;118(4):1654-9. doi: 10.1542/peds.2005-2463. PMID 17015558
- [Result] Walsh M, Laptook A, Kazzi SN, Engle WA, Yao Q, Rasmussen M, Buchter S, Heldt G, Rhine W, Higgins R, Poole K; National Institute of Child Health and Human Development Neonatal Research Network. A cluster-randomized trial of benchmarking and multimodal quality improvement to improve rates of survival free of bronchopulmonary dysplasia for infants with birth weights of less than 1250 grams. Pediatrics. 2007 May;119(5):876-90. doi: 10.1542/peds.2006-2656. PMID 17473087
- [Result] Walsh M, Engle W, Laptook A, Kazzi SN, Buchter S, Rasmussen M, Yao Q; National Institute of Child Health and Human Development Neonatal Research Network. Oxygen delivery through nasal cannulae to preterm infants: can practice be improved? Pediatrics. 2005 Oct;116(4):857-61. doi: 10.1542/peds.2004-2411. PMID 16199694
- [Result] Wilson-Costello D, Walsh MC, Langer JC, Guillet R, Laptook AR, Stoll BJ, Shankaran S, Finer NN, Van Meurs KP, Engle WA, Das A; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Impact of postnatal corticosteroid use on neurodevelopment at 18 to 22 months' adjusted age: effects of dose, timing, and risk of bronchopulmonary dysplasia in extremely low birth weight infants. Pediatrics. 2009 Mar;123(3):e430-7. doi: 10.1542/peds.2008-1928. Epub 2009 Feb 9. PMID 19204058
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/